CLINICAL TRIAL: NCT02786134
Title: Coronary Flow Reserve to Assess Cardiovascular Inflammation (CIRT-CFR)
Acronym: CIRT-CFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Ottawa Heart Institute Research Corporation (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Marcelo F. Di Carli, MD, FACC, Chief of Nuclear Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2013P002186
Record Dates: First submitted 2016-05-20; First posted 2016-05-30 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Coronary Heart Disease; Metabolic Syndrome; Diabetes Mellitus
MeSH Terms: conditions — Coronary Disease; Metabolic Syndrome; Diabetes Mellitus | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: The CIRT-CFR study is a sub-study based off the main CIRT trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- low-dose methotrexate (LDM) (Experimental): Patients willing to participate in CIRT will be asked to enroll into the sub-study and may sign the CIRT-CFR informed consent at any point between signing the parent CIRT informed consent and completing the parent CIRT randomization visit (Visit 4). After giving informed consent for the ancillary CIRT-CFR, patients will undergo the baseline rest/dipyridamole stress PET scan along with echocardiography. The final PET scan and echocardiogram will occur at approximately 12 months after randomization.
  Interventions: Radiation: PET scan; Radiation: Echocardiogram
- placebo (Experimental): Patients willing to participate in CIRT will be asked to enroll into the sub-study and may sign the CIRT-CFR informed consent at any point between signing the parent CIRT informed consent and completing the parent CIRT randomization visit (Visit 4). After giving informed consent for the ancillary CIRT-CFR, patients will undergo the baseline rest/dypridamole stress PET scan along with echocardiography. The final PET scan and echocardiogram will occur at approximately 12 months after randomization.
  Interventions: Radiation: PET scan; Radiation: Echocardiogram

INTERVENTIONS:
Radiation: PET scan — A cardiac PET scan will be performed at baseline (main CIRT trial randomization) and at 12-months.
Radiation: Echocardiogram — An echocardiogram will be performed at baseline (main CIRT trial randomization) and at 12-months.

SUMMARY:
Coronary flow reserve (CFR, calculated as the ratio of hyperemic over rest myocardial blood flow) is emerging as a powerful quantitative prognostic imaging marker of clinical cardiovascular risk. CFR provides a robust and reproducible clinical measure of the integrated hemodynamic effects of epicardial coronary artery disease (CAD), diffuse atherosclerosis, and microvascular dysfunction on myocardial tissue perfusion. Inflammation is a key mediator of this constellation of abnormalities, affecting the entire coronary vasculature, but no clinical trial to date has shown that directly reducing inflammation lowers cardiovascular event rates. As such, the recently launched Cardiovascular Inflammation Reduction Trial (CIRT) provides a unique opportunity for mechanistic investigation of the impact of anti-inflammatory therapy on changes in CFR as a reflection of coronary vascular dysfunction, which may precede clinical outcomes, particularly in patients at high-risk of events. The investigators are ideally positioned to examine the impact of inflammation on CFR, having extensive experience in both the quantitation of CFR using clinically-integrated dynamic positron emission tomography (PET) and the ability to assess its association with cardiovascular outcomes. The central hypothesis of this ancillary proposal, CIRT-CFR, is that reducing systemic inflammation using low-dose methotrexate (LDM) will, compared to placebo, quantitatively improve myocardial blood flow and coronary flow reserve as measured by PET over one year, in stable CAD patients with type 2 diabetes or metabolic syndrome enrolled in CIRT. In so doing, improvement in coronary vasoreactivity, endothelial function, and tissue perfusion may have beneficial effects on myocardial mechanics, left ventricular deformation and function and, ultimately, symptoms and prognosis.

DETAILED DESCRIPTION:
Randomization and double-blind study treatment period to either placebo or LDM (1:1) of willing and eligible patients will occur at the end of the open label run-in phase per the parent CIRT protocol, and will be stratified by time since the qualifying event (< 6 or ≥ 6 months from the date of MI or most recent angiogram), type of event (MI or multivessel CAD), presence of either type 2 DM or metabolic syndrome, and site, which will ensure balance in the proposed study. Patients willing to participate in CIRT will be asked to enroll into the sub-study and may sign the CIRT-CFR informed consent at any point between signing the parent CIRT informed consent and completing the parent CIRT randomization visit (Visit 4). After giving informed consent for the ancillary CIRT-CFR, patients will undergo the baseline PET scan along with echocardiography at any point between the parent CIRT post run-in visit (Visit 3) and up to 4 weeks after randomization (Visit 4).

Imaging will be performed at the 3 imaging centers (BWH, OHI, and UAB). To minimize participant and site burden, only a baseline and single follow-up imaging time point will be pursued. Imaging tests (PET and echo) will be scheduled on the same day for patient convenience if possible, and no more than one week apart. "Baseline" study visit imaging will follow the open label run-in period of the parent trial to enhance long-term compliance and eliminate risk of radiation exposure for any individuals with immediate intolerance to the LDM study protocol. The imaging tests proposed are non-invasive, routinely performed, and historically well tolerated by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at screening;
2. Documented past history of MI OR past evidence of multivessel CAD by angiography, completed any planned coronary revascularization associated with a qualifying event at least 60 days prior to enrollment, and clinically stable for ≥60 days prior to enrollment; qualifying prior MI must be documented either by hospital records, evidence on current ECG of Q waves in 2 contiguous leads, and/or an imaging test demonstrating wall motion abnormality or scar; qualifying evidence of multivessel CAD by angiography must be documented by CAD in at least two major epicardial vessels defined either as the presence of a stent, a coronary artery bypass graft, or an angiographic lesion of 60% or greater (left main CAD that has been revascularized with a stent or bypass graft will qualify as multivessel disease, as will the presence of a 50% or greater isolated left main stenosis);
3. History of type 2 DM or metabolic syndrome (meeting 2004 AHA/NHLBI definition*) at time of study enrollment; *includes any 3 of the following 5 diagnostic criteria: waist circumference ≥ 102 cm in men or 88 cm in women; triglycerides ≥ 150 mg/dl or on drug treatment for elevated triglycerides; high-density lipoprotein cholesterol (HDL-C)< 40 mg/dL in men or < 50 mg/dL in women or on drug treatment for reduced HDL-C; systolic blood pressure ≥ 130 mm Hg or diastolic blood pressure ≥ 85 mm Hg or on drug treatment for hypertension; and elevated fasting glucose ≥ 100 mg/dL or on drug treatment for elevated glucose.
4. Willingness to participate as evidenced by signing the CIRT and CIRT-CFR informed consent.

Exclusion criteria:

1. Prior history of chronic infectious disease, tuberculosis, or severe fungal disease; chronic hepatitis B or C infection; renal insufficiency; interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis; known chronic pericardial effusion, pleural effusion, or ascites; chronic liver disease; myeloproliferative disorders in the past 5 years; non-basal cell malignancy or treated lymphoproliferative disease within the past 5 years; known HIV positive; life expectancy of <3 years;
2. Chronic inflammatory condition such as lupus or rheumatoid arthritis, ulcerative colitis or Crohn's disease
3. White blood cell count <3,500/ul, hematocrit < 32 percent, or platelet count < 75,000/ul
4. Liver transaminase levels (AST or ALT) >upper limit of normal (ULN) or albumin < the lower limit of normal (LLN);
5. Creatinine clearance < 40 ml/min as estimated with the Cockroft-Gault equation;
6. History of alcohol abuse or unwillingness to limit alcohol consumption to less than 4 drinks per week
7. Women of child bearing potential, even if they are currently using contraception, and women intending to breastfeed.
8. Men who plan to father children during the study period or who are unwilling to use effective forms of contraception.
9. Requirement for use of drugs that alter folate metabolism (trimethoprim/sulfamethoxazol) or reduce tubular excretion (probenecid) or known allergies to antibiotics making avoidance of trimethoprim impossible;
10. Current indication for methotrexate therapy;
11. Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers (see Exclusionary Medication List in Manual of Operations). Eligible study participants will be encouraged to have up to date pneumococcal and influenza vaccinations as recommended based on their age and underlying medical conditions.
12. Chest X-ray evidence in the past 12 months of interstitial pneumonitis, bronchiectasis, or pulmonary fibrosis. For participants who do not have a chest X-ray in the prior 12 months, a chest X-ray will be obtained at baseline as part of the study protocol.
13. New York Heart Association Class IV congestive heart failure.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Taqueti VR, Shah AM, Everett BM, Pradhan AD, Piazza G, Bibbo C, Hainer J, Morgan V, Carolina do A H de Souza A, Skali H, Blankstein R, Dorbala S, Goldhaber SZ, Le May MR, Chow BJW, deKemp RA, Hage FG, Beanlands RS, Libby P, Glynn RJ, Solomon SD, Ridker PM, Di Carli MF. Coronary Flow Reserve, Inflammation, and Myocardial Strain: The CIRT-CFR Trial. JACC Basic Transl Sci. 2022 Dec 21;8(2):141-151. doi: 10.1016/j.jacbts.2022.08.009. eCollection 2023 Feb. PMID 36908662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Dose Methotrexate (LDM) | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose Methotrexate (LDM) | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 16 | 28
  >=65 years | 13 | 9 | 22
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 66 [61 to 73] | 63 [57 to 68] | 65 [59 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 25 | 22 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 23 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Myocardial Blood Flow in Response to Vasodilator
Description: Change (from baseline) in global coronary flow reserve in response to vasodilator as measured by PET imaging at baseline and at one year
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percentage change in CFR
Arm/Group | Low-Dose Methotrexate (LDM) | Placebo
Number analyzed (Participants) | 25 | 25
percentage change in CFR | 0.05 [-0.192 to 0.288] | -0.145 [-0.429 to 0.117]

ADVERSE EVENTS:
Time Frame: 1 year
Description: The adverse definitions match those listed on clincaltrials.gov.
Arm/Group | Low-Dose Methotrexate (LDM) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 2/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Methotrexate (LDM) (N=25) | Placebo (N=25)
Shortness of Breath during PET scan (Cardiac disorders) | 0 (0) | 2 (2)
Headache during PET scan (Cardiac disorders) | 0 (0) | 1 (2)
Chest Pain during PET scan (Cardiac disorders) | 2 (3) | 0 (0)
Swelling at IV site (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Developed atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT02786134/Prot_SAP_000.pdf